CLINICAL TRIAL: NCT01588990
Title: An Australian Translational Study to Evaluate the Prognostic Role of Inflammatory Markers in Patients With Metastatic Colorectal Cancer Treated With Bevacizumab (Avastin™)
Brief Title: A Translational Study of Bevacizumab in Participants With Metastatic Colorectal Cancer
Acronym: ASCENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25753
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Bevacizumab; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab: Phase A and Phase B (Experimental): The trial will consist of 2 phases of treatment. Phase A: Participants will receive bevacizumab 7.5 mg/kg intravenous (IV) infusion on Day 1 every 3 weeks in combination with XELOX (capecitabine and oxaliplatin) or bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with mFOLFOX6 (oxaliplatin, leucovorin, and 5-fluouracil) until first disease progression or occurrence of unmanageable toxicity. Phase B: Upon documented first disease progression, participants will continue receiving bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with FOLFIRI (irinotecan, leucovorin, and 5-fluouracil) until second disease progression or occurrence of unmanageable toxicity. Phase B treatment should commence within 4 weeks of the date of documented first disease progression.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab; Drug: Leucovorin; Drug: 5-Fluouracil; Drug: Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin — Participants will receive oxaliplatin 85 milligrams per square meter (mg/m^2) IV infusion on Day 1 of every 2 weeks cycle during alternative Phase A treatment or 130 mg/m^2 on Day 1 of every 3 weeks cycle during Phase A treatment.
Drug: Capecitabine — Participants will receive capecitabine 1000 mg/m^2 per oral (PO) twice daily on Days 1-14 of 3 weeks cycle during Phase A treatment.
Drug: Bevacizumab — Participants will receive 7.5 mg/kg IV infusion on Day 1 every 3 weeks (Phase A treatment) or 5 mg/kg IV on Day 1 every 2 weeks (Alternative Phase A treatment and Phase B).
  Other Names: Avastin, RO4876646
Drug: Leucovorin — Participants will receive leucovorin 400 mg/m^2 IV on Day 1 every 2 weeks (Alternative Phase A treatment and Phase B). Investigators may elect to chose low dose of leucovorin (either 20 mg/m^2 or 50 mg total dose).
Drug: 5-Fluouracil — Participants will receive 5-fluouracil loading dose of 400 mg/m^2 IV on Day 1 followed by 2400 mg/m^2 continuous IV infusion over 46 hours Day 1 (Alternative Phase A treatment and Phase B).
Drug: Irinotecan — Participants will receive irinotecan 180 mg/m^2 IV on Day 1 every 2 weeks during Phase B treatment.

SUMMARY:
This open-label, prospective, single-arm, multicenter study will evaluate the relationship of the markers of inflammation and progression-free survival (PFS) in participants with previously untreated metastatic colorectal cancer. The study consists of two phases: Phase A treatment: oral capecitabine plus infusional oxaliplatin (XELOX) plus bevacizumab, or modified infusional 5-fluorouracil (5-FU), leucovorin (LV) and oxaliplatin (mFOLFOX6) plus bevacizmab administered until first disease progression. Participants will then continue with Phase B treatment: infusional 5-FU, LV and irinotecan (FOLFIRI) plus bevacizumab until second disease progression. The anticipated time on study treatment is 4 years.

ELIGIBILITY:
Inclusion Criteria:

For resected primary tumor participants, and participants with primary tumor in situ:

* Previously untreated metastatic colorectal cancer and not a candidate for curative resection
* World Health Organization (WHO) performance status of 0-1
* Life expectancy of greater than or equal to (>/=) 3 months
* Eligible for XELOX, mFOLFOX6, FOLFIRI and bevacizumab treatment in accordance with local standards of care and pharmaceutical benefits scheme guidelines

Additional inclusion criteria for participants with primary tumor in situ:

* Intact primary tumor of the colon or the rectum not requiring surgical intervention prior to study start
* Minimal or asymptomatic primary tumor

Exclusion Criteria:

Resected primary tumor participants, and participants with primary tumor in situ:

* Previous chemotherapy for metastatic colorectal cancer
* Previous neoadjuvant or adjuvant chemotherapy less than 6 months prior to study start
* Radiotherapy within 28 days prior to enrollment or not recovered from a radiotherapy
* History of non-colorectal cancer (participants are eligible if disease-free for >/=5 years and the risk of recurrence is deemed low)
* Presence of active inflammatory bowel disease
* History of gastrointestinal perforations
* Peritoneal disease
* History of significant bleeding event
* Significant vascular disease
* Peripheral arterial thrombosis or other thrombotic event within 6 months before study start

Additional exclusion criteria for participants with primary tumor in situ:

* Prior endoscopic management of the current tumor
* Acute diverticulitis
* Presence of intra-abdominal abscess
* Active gastroduodenal ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Australia (17):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent'S Hospital; Clinical Oncology, Darlinghurst, New South Wales
  - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Royal North Shore Hospital; Department of Medical Oncology, St Leonards, New South Wales
  - Sydney Adventist Hospital; Clinical Trial Unit, Sydney, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - The Townsville Hospital; Townsville Cancer Centre, Townsville, Queensland
  - Lyell McEwin Hospital; Oncology Clinical Trials, Chemotherapy Day Unit, Elizabeth Vale, South Australia
  - Calvary North Adelaide; North Adeliade Oncology Centre, North Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
  - Sunshine Hospital; Oncology Research, St Albans, Victoria
  - St John of God Murdoch Hospital; Oncology West, Murdoch, Western Australia
  - St John of God Hospital; Bendat Cancer Centre, Subiaco, Western Australia

REFERENCES:
- [Derived] Clarke SJ, Burge M, Feeney K, Gibbs P, Jones K, Marx G, Molloy MP, Price T, Reece WHH, Segelov E, Tebbutt NC. The prognostic role of inflammatory markers in patients with metastatic colorectal cancer treated with bevacizumab: A translational study [ASCENT]. PLoS One. 2020 Mar 6;15(3):e0229900. doi: 10.1371/journal.pone.0229900. eCollection 2020. PMID 32142532
- [Derived] Clarke S, Burge M, Cordwell C, Gibbs P, Reece W, Tebbutt N. An Australian translational study to evaluate the prognostic role of inflammatory markers in patients with metastatic ColorEctal caNcer Treated with bevacizumab (Avastin) [ASCENT]. BMC Cancer. 2013 Mar 15;13:120. doi: 10.1186/1471-2407-13-120. PMID 23497305

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Phase A and Phase B: The trial consisted of 2 phases of treatment. Phase A: Participants received bevacizumab 7.5 mg/kg IV on Day 1 every 3 weeks in combination with XELOX (oral capecitabine 1000 mg/m^2 twice daily Days 1-14, oxaliplatin 130 mg/m^2 IV Day 1) or bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with mFOLFOX6 (oxaliplatin 85 mg/m^2 IV Day 1, leucovorin 400 mg/m^2 IV Day 1, 5-fluouracil 400 mg/m^2 IV loading dose then 2400 mg/m^2 continuous IV infusion over 46 hours Day 1) until first disease progression or occurrence of unmanageable toxicity. Phase B: Upon documented first disease progression, participants continued receiving bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with FOLFIRI (irinotecan 180 mg/m^2 IV Day 1, leucovorin and 5-fluouracil [same regimen as of mFOLFOX6]) until second disease progression or occurrence of unmanageable toxicity. Phase B treatment had to commence within 4 weeks of the date of documented first disease progression.
Period: Phase A
Arm/Group | Bevacizumab: Phase A and Phase B
Started | 128
Completed | 58 (A total of 58 participants had disease progression in Phase A and ended Phase A.)
Not Completed | 70
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 11
Not completed — Other | 14
Not completed — Lost to Follow-up | 1
Not completed — Death | 5
Not completed — Adverse Event | 28
Not completed — Still on therapy at end of study | 6
Period: Phase B
Arm/Group | Bevacizumab: Phase A and Phase B
Started | 53 (Of 58 participants who had documented disease progression in Phase A, 53 entered in Phase B.)
Completed | 37 (A total of 37 participants had disease progression in Phase B and ended Phase B.)
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Still on therapy at end of study | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 4
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of bevacizumab.
Groups:
- Bevacizumab: Phase A and Phase B: The trial consisted of 2 phases of treatment. Phase A: Participants received bevacizumab 7.5 mg/kg intravenously (IV) on Day 1 every 3 weeks in combination with XELOX (oral capecitabine 1000 mg/m^2 twice daily Days 1-14, oxaliplatin 130 mg/m^2 IV Day 1) or bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with mFOLFOX6 (oxaliplatin 85 mg/m^2 IV Day 1, leucovorin 400 mg/m^2 IV Day 1, 5-fluouracil 400 mg/m^2 IV loading dose then 2400 mg/m^2 continuous IV infusion over 46 hours Day 1) until first disease progression or occurrence of unmanageable toxicity. Phase B: Upon documented first disease progression, participants continued receiving bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with FOLFIRI (irinotecan 180 mg/m^2 IV Day 1, leucovorin and 5-fluouracil [same regimen as of mFOLFOX6]) until second disease progression or occurrence of unmanageable toxicity. Phase B treatment had to commence within 4 weeks of the date of documented first disease progression.
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Association Between Neutrophil to Lymphocyte Ratio (NLR) [NLR ≤5 Versus NLR >5] and Progression-Free Survival (PFS) as Assessed by Hazard Ratio
Description: NLR was calculated from the laboratory values as the ratio of Neutrophils to Lymphocytes. PFS was defined as the time from the start of initial treatment to documentation of first disease progression or death from any cause, whichever occurred first. Disease progression was determined according to standard practice based on radiological, biochemical (carcinoembryonic antigen [CEA]) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. The association between NLR (NLR less than or equal to [≤] 5 vs greater than [>] 5) and PFS was reported as hazard ratio.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 127
hazard ratio | 1.4 [0.9 to 2.2]
Statistical Analysis 1: Comparison: Bevacizumab: Phase A and Phase B; Test type: Superiority or Other; p = 0.101, Cox Proportional Hazards Model

2. Secondary Outcome: PFS Until First Disease Progression as Assessed by the Investigator Based on Routine Clinical Practice: Phase A
Description: PFS until first progression was defined as the time from the start of initial treatment to documentation of first disease progression or death from any cause, whichever occurred first. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: Baseline up to first disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab: Phase A: In Phase A, participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) IV on Day 1 every 3 weeks in combination with XELOX (oral capecitabine 1000 milligrams per square meter [mg/m^2] twice daily Days 1-14, oxaliplatin 130 mg/m^2 IV Day 1) or bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with mFOLFOX6 (oxaliplatin 85 mg/m^2 IV Day 1, leucovorin 400 mg/m^2 IV Day 1, 5-fluouracil 400 mg/m^2 IV loading dose then 2400 mg/m^2 continuous IV infusion over 46 hours Day 1) until first disease progression or occurrence of unmanageable toxicity.
Arm/Group | Bevacizumab: Phase A
Number analyzed (Participants) | 128
months | 9.2 [7.9 to 10.8]

3. Secondary Outcome: PFS Until Second Disease Progression as Assessed by the Investigator Based on Routine Clinical Practice: Phase B
Description: PFS in Phase B (PFS-B) was defined as the time from the start of Phase B treatment to documentation of second disease progression or death from any cause, whichever occurred first. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: From the start of Phase B treatment to disease progression, death or end of study (up to 4 years)
Population: Phase B FAS population included participants who received at least 1 dose of bevacizumab in Phase B.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab: Phase B: Upon documented first disease progression in Phase A, participants continued receiving bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with FOLFIRI (irinotecan 180 mg/m^2 IV Day 1, leucovorin 400 mg/m^2 IV Day 1, and 5-fluouracil 400 mg/m^2 IV loading dose then 2400 mg/m^2 continuous IV infusion over 46 hours Day 1) in Phase B until second disease progression or occurrence of unmanageable toxicity. Phase B treatment had to commence within 4 weeks of the date of documented first disease progression.
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
months | 6.7 [3.0 to 8.2]

4. Secondary Outcome: Time to Failure of Strategy (TFS): Overall
Description: TFS was defined as time from the start of initial treatment to documentation of first disease progression without entering Phase B, or second disease progression having entered Phase B. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. Kaplan-Meier methodology was used to estimate TFS.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
months | 14.8 [13.1 to 19.4]

5. Secondary Outcome: Duration of Disease Control (DDC) as Assessed by the Investigator Based on Routine Clinical Practice: Overall
Description: DDC was defined as PFS + PFS-B. In cases where a participant did not enter Phase B, then DDC was defined as PFS. PFS was defined as time from start of initial treatment to documentation of first disease progression or death from any cause, whichever occurred first. PFS-B was time from start of Phase B treatment to documentation of second disease progression or death from any cause, whichever occurred first. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. Kaplan-Meier methodology was used to estimate DDC.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
months | 14.0 [10.8 to 16.6]

6. Secondary Outcome: Overall Survival (OS) From the Start of Treatment to Study Completion: Overall
Description: OS was defined as the time from the start of initial treatment to the date of death, regardless of the cause of death. Kaplan-Meier methodology was used to estimate OS.
Time Frame: Baseline until death or end of study (up to 4 years)
Population: FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
months | 25.0 [19.2 to 29.7]

7. Secondary Outcome: Survival Beyond First Disease Progression: Overall
Description: Survival beyond first progression was defined as the time from the date of first disease progression to death due to any cause. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as any of the following: an unequivocal and clinically meaningful increase in the size of known tumors, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. Kaplan-Meier methodology was used to estimate survival beyond first disease progression.
Time Frame: Baseline until death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 101
months | 12.6 [8.8 to 15.9]

8. Secondary Outcome: OS: Phase B
Description: Overall Survival in Phase B was defined as the time from the start of treatment in Phase B to death due to any cause. Kaplan-Meier methodology was used to estimate OS.
Time Frame: From the start of Phase B treatment death or end of study (up to 4 years)
Population: Phase B FAS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
months | 14.9 [8.2 to 17.5]

9. Secondary Outcome: Percentage of Participants With Confirmed Complete or Partial Response as Assessed by the Investigator Based on Routine Clinical Practice: Phase A
Description: Percentage of participants with best overall response of confirmed complete response or partial response based on the investigator assessment of the response as per routine clinical practice was reported. The confirmation of response must be no less than 4 weeks after initial assessment.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab: Phase A: In Phase A, participants received bevacizumab 7.5 mg/kg IV on Day 1 every 3 weeks in combination with XELOX (oral capecitabine 1000 mg/m^2 twice daily Days 1-14, oxaliplatin 130 mg/m^2 IV Day 1) or bevacizumab 5 mg/kg IV on Day 1 every 2 weeks in combination with mFOLFOX6 (oxaliplatin 85 mg/m^2 IV Day 1, leucovorin 400 mg/m^2 IV Day 1, 5-fluouracil 400 mg/m^2 IV loading dose then 2400 mg/m^2 continuous IV infusion over 46 hours Day 1) until first disease progression or occurrence of unmanageable toxicity.
Arm/Group | Bevacizumab: Phase A
Number analyzed (Participants) | 128
percentage of participants
  Complete response | 3.1
  Partial response | 8.6

10. Secondary Outcome: Percentage of Participants With Confirmed Complete or Partial Response as Assessed by the Investigator Based on Routine Clinical Practice: Phase B
Description: as for outcome 9
Time Frame: From the start of Phase B treatment to disease progression, death or end of study (up to 4 years)
Population: Phase B FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
percentage of participants
  Complete response | 0
  Partial response | 0

11. Secondary Outcome: Percentage of Participants With Confirmed Complete or Partial Response as Assessed by the Investigator Based on Routine Clinical Practice: Overall
Description: as for outcome 9
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
percentage of participants
  Complete response | 3.1
  Partial response | 8.6

12. Secondary Outcome: Percentage of Participants Who Underwent Liver Resection: Overall
Description: The results include percentage of participants who underwent potentially curative liver resection.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 128
percentage of participants | 1.6

13. Secondary Outcome: Association Between NLR (NLR ≤5 Versus NLR >5) and OS as Assessed by Hazard Ratio
Description: NLR was calculated from the laboratory values as the ratio of Neutrophils to Lymphocytes. OS was defined as the time from the start of initial treatment to the date of death, regardless of the cause of death. The association between NLR (NLR ≤ 5 vs > 5) and OS was reported as hazard ratio.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 127
hazard ratio | 1.6 [1.0 to 2.7]
Statistical Analysis 1: Comparison: Bevacizumab: Phase A and Phase B; Test type: Superiority or Other; p = 0.052, Cox Proportional Hazards Model

14. Secondary Outcome: Association Between NLR Normalization (First NLR Post-Baseline ≤5 Versus NLR >5) and PFS as Assessed by Hazard Ratio
Description: NLR was calculated from laboratory values as ratio of Neutrophils to Lymphocytes. NLR normalization was assessed by adding first post-baseline measurement of NLR to the primary model. This is equivalent to testing whether first change in NLR is significantly associated with outcome. PFS was defined as time from start of initial treatment to documentation of first disease progression or death from any cause. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was defined as: an unequivocal and clinically meaningful increase in size of known tumors, appearance of ≥1 new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration.The association between NLR normalization (first NLR post-baseline ≤5 vs >5) and PFS was reported as hazard ratio.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 127
hazard ratio | 0.9 [0.5 to 1.8]
Statistical Analysis 1: Comparison: Bevacizumab: Phase A and Phase B; Test type: Superiority or Other; p = 0.797, Cox Proportional Hazards Model

15. Secondary Outcome: Association Between Longitudinal NLR (Longitudinal NLR ≤5 Versus NLR >5) and PFS as Assessed by Hazard Ratio
Description: NLR was calculated from the laboratory values as the ratio of Neutrophils to Lymphocytes. Longitudinal NLR was assessed by treating the NLR measurements taken over the time-course of treatment as a time-dependent covariate. PFS was defined as time from the start of initial treatment to documentation of first disease progression or death from any cause, whichever occurred first. Disease progression was determined according to standard practice based on radiological, biochemical (CEA) or clinical factors. Determination of disease progression was to be unequivocal and was defined as: an unequivocal and clinically meaningful increase in size of known tumors, appearance of one or more new lesions, death due to disease without prior objective documentation of progression, elevated CEA accompanied by other radiological or clinical evidence of progression, or symptomatic deterioration. The association between longitudinal NLR (longitudinal NLR ≤5 vs N>5) and PFS was reported as hazard ratio.
Time Frame: Baseline up to disease progression, death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 127
hazard ratio | 1.3 [0.9 to 1.9]
Statistical Analysis 1: Comparison: Bevacizumab: Phase A and Phase B; Test type: Superiority or Other; p = 0.188, Cox Proportional Hazards Model

16. Secondary Outcome: Association Between Longitudinal NLR (Longitudinal NLR ≤5 Versus NLR >5) and OS as Assessed by Hazard Ratio
Description: NLR was calculated from the laboratory values as the ratio of Neutrophils to Lymphocytes. Longitudinal NLR was assessed by treating the NLR measurements taken over the time-course of treatment as a time-dependent covariate. OS was defined as the time from the start of initial treatment to the date of death, regardless of the cause of death. The association between longitudinal NLR (longitudinal NLR ≤5 vs NLR >5) and OS was reported as hazard ratio.
Time Frame: Baseline up to death or end of study (up to 4 years)
Population: FAS population. "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Bevacizumab: Phase A and Phase B
Number analyzed (Participants) | 127
hazard ratio | 2.2 [1.2 to 4.0]
Statistical Analysis 1: Comparison: Bevacizumab: Phase A and Phase B; Test type: Superiority or Other; p = 0.016, Cox Proportional Hazards Model

17. Secondary Outcome: European Quality of Life 5-Dimension (EuroQol-5D) Utility Score: Phase A
Description: EQ-5D is a standardized generic preference based health related quality of life instrument. It records how one's health is "today" and consists of a descriptive system. The descriptive system is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension on the EQ-5D involves a 3-point response scale which indicates the level of impairment (level 1 = no problem; level 2 = some or moderate problem[s] and level 3 = unable, or extreme problems). Level of problem reported in each EQ-5D dimension determines a unique health state which is converted into a weighted health state index by applying scores from EQ-5D preference weights elicited from general population samples. This generates a unique description of the subjects' health status, which is valued between 0 (representing death) and 1 (representing perfect health). Higher the score, the better the quality of life.
Time Frame: Baseline, every 8-9 weeks thereafter, end of treatment (EOT) (30 days after disease progression [up to 4 years]), survival follow-up 12-weekly visits (up to 4 years) [Detailed time points are presented in the category titles]
Population: FAS population. "Number Analyzed" = participants who were evaluable at the specified time point for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase A
Number analyzed (Participants) | 128
units on a scale
  Phase A Baseline: number analyzed (Participants) | 127
  Phase A Baseline | 0.830 (0.1590)
  Phase A Visit 2 (Weeks 8-9): number analyzed (Participants) | 100
  Phase A Visit 2 (Weeks 8-9) | 0.857 (0.1392)
  Phase A Visit 3 (Weeks 16-17): number analyzed (Participants) | 79
  Phase A Visit 3 (Weeks 16-17) | 0.865 (0.1074)
  Phase A Visit 4 (Weeks 24-25): number analyzed (Participants) | 62
  Phase A Visit 4 (Weeks 24-25) | 0.853 (0.1206)
  Phase A Visit 5 (Weeks 32-33): number analyzed (Participants) | 42
  Phase A Visit 5 (Weeks 32-33) | 0.869 (0.1381)
  Phase A Visit 6 (Weeks 40-41): number analyzed (Participants) | 30
  Phase A Visit 6 (Weeks 40-41) | 0.892 (0.1013)
  Phase A Visit 7 (Weeks 48-49): number analyzed (Participants) | 23
  Phase A Visit 7 (Weeks 48-49) | 0.872 (0.1332)
  Phase A Visit 8 (Weeks 56-57): number analyzed (Participants) | 18
  Phase A Visit 8 (Weeks 56-57) | 0.881 (0.1058)
  Phase A Visit 9 (Weeks 64-65): number analyzed (Participants) | 19
  Phase A Visit 9 (Weeks 64-65) | 0.894 (0.1081)
  Phase A Visit 10 (Weeks 72-73): number analyzed (Participants) | 15
  Phase A Visit 10 (Weeks 72-73) | 0.843 (0.1466)
  Phase A Visit 11 (Weeks 80-81): number analyzed (Participants) | 14
  Phase A Visit 11 (Weeks 80-81) | 0.898 (0.0952)
  Phase A Visit 12 (Weeks 88-89): number analyzed (Participants) | 14
  Phase A Visit 12 (Weeks 88-89) | 0.915 (0.1033)
  Phase A Visit 13 (Weeks 96-97): number analyzed (Participants) | 12
  Phase A Visit 13 (Weeks 96-97) | 0.844 (0.1463)
  Phase A Visit 14 (Weeks 104-105): number analyzed (Participants) | 12
  Phase A Visit 14 (Weeks 104-105) | 0.899 (0.1398)
  Phase A Visit 15 (Weeks 112-113): number analyzed (Participants) | 10
  Phase A Visit 15 (Weeks 112-113) | 0.878 (0.0861)
  Phase A Visit 16 (Weeks 120-121): number analyzed (Participants) | 8
  Phase A Visit 16 (Weeks 120-121) | 0.899 (0.0852)
  Phase A Visit 17 (Weeks 128-129): number analyzed (Participants) | 10
  Phase A Visit 17 (Weeks 128-129) | 0.873 (0.1734)
  Phase A Visit 18 (Weeks 136-137): number analyzed (Participants) | 9
  Phase A Visit 18 (Weeks 136-137) | 0.909 (0.0876)
  Phase A Visit 19 (Weeks 144-145): number analyzed (Participants) | 7
  Phase A Visit 19 (Weeks 144-145) | 0.947 (0.0914)
  Phase A Visit 20 (Weeks 152-153): number analyzed (Participants) | 7
  Phase A Visit 20 (Weeks 152-153) | 0.852 (0.0718)
  Phase A Visit 21 (Weeks 160-161): number analyzed (Participants) | 3
  Phase A Visit 21 (Weeks 160-161) | 0.933 (0.1156)
  Phase A Visit 22 (Weeks 168-169): number analyzed (Participants) | 2
  Phase A Visit 22 (Weeks 168-169) | 0.813 (0.0193)
  Phase A Visit 23 (Weeks 176-177): number analyzed (Participants) | 2
  Phase A Visit 23 (Weeks 176-177) | 0.900 (0.1416)
  Phase A EOT Visit (up to 4 years): number analyzed (Participants) | 78
  Phase A EOT Visit (up to 4 years) | 0.817 (0.1423)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 10
  Survival Follow-Up 1 (up to 4 years) | 0.768 (0.1414)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 2 (up to 4 years) | 0.901 (0.0860)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 2
  Survival Follow-Up 3 (up to 4 years) | 0.819 (0.0583)
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 0.843
  Survival Follow-Up 5 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 5 (up to 4 years) | 1.000
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 6 (up to 4 years) | 0.835 (0.0229)
  Survival Follow-Up 7 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 7 (up to 4 years) | 0.816

18. Secondary Outcome: EuroQol-5D Utility Score: Phase B
Description: as for outcome 17
Time Frame: Baseline, every 8-9 weeks thereafter, EOT (30 days after disease progression [up to 4 years]), survival follow-up 12-weekly visits (up to 4 years) [Detailed time points are presented in the category titles]
Population: Phase B FAS population. "Number Analyzed" = participants who were evaluable at the specified time point for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
units on a scale
  Phase B Baseline | 0.814 (0.1566)
  Phase B Visit 2 (up to 4 years): number analyzed (Participants) | 32
  Phase B Visit 2 (up to 4 years) | 0.859 (0.1376)
  Phase B Visit 3 (up to 4 years): number analyzed (Participants) | 25
  Phase B Visit 3 (up to 4 years) | 0.894 (0.1108)
  Phase B Visit 4 (up to 4 years): number analyzed (Participants) | 20
  Phase B Visit 4 (up to 4 years) | 0.897 (0.1012)
  Phase B Visit 5 (up to 4 years): number analyzed (Participants) | 13
  Phase B Visit 5 (up to 4 years) | 0.866 (0.1299)
  Phase B Visit 6 (up to 4 years): number analyzed (Participants) | 12
  Phase B Visit 6 (up to 4 years) | 0.837 (0.1710)
  Phase B Visit 7 (up to 4 years): number analyzed (Participants) | 6
  Phase B Visit 7 (up to 4 years) | 0.876 (0.0986)
  Phase B Visit 8 (up to 4 years): number analyzed (Participants) | 3
  Phase B Visit 8 (up to 4 years) | 0.874 (0.1141)
  Phase B Visit 9 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 9 (up to 4 years) | 0.908 (0.1299)
  Phase B Visit 10 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 10 (up to 4 years) | 0.811 (0.0466)
  Phase B Visit 11 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 11 (up to 4 years) | 0.806 (0.0539)
  Phase B Visit 12 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 12 (up to 4 years) | 0.844
  Phase B Visit 13 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 13 (up to 4 years) | 1.000
  Phase B Visit 14 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 14 (up to 4 years) | 1.000
  Phase B Visit 15 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 15 (up to 4 years) | 0.844
  Phase B Visit 16 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 16 (up to 4 years) | 0.833
  Phase B Visit 17 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 17 (up to 4 years) | 0.844
  Phase B Visit 18 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 18 (up to 4 years) | 0.833
  Phase B Visit 19 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 19 (up to 4 years) | 0.827
  Phase B Visit 20 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 20 (up to 4 years) | 0.816
  Phase B Visit 21 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 21 (up to 4 years) | 0.844
  Phase B Visit 22 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 22 (up to 4 years) | 0.844
  Phase B Visit 23 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 23 (up to 4 years) | 0.827
  Phase B Visit 24 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 24 (up to 4 years) | 0.844
  Phase B EOT Visit (up to 4 years): number analyzed (Participants) | 31
  Phase B EOT Visit (up to 4 years) | 0.809 (0.1585)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 1 (up to 4 years) | 0.740 (0.1035)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 4
  Survival Follow-Up 2 (up to 4 years) | 0.772 (0.0782)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 3 (up to 4 years) | 0.827
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 0.827
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 6 (up to 4 years) | 1.000

19. Secondary Outcome: Assessment of Quality of Life - Eight Dimensions (AQoL-8D) Global Utility Score: Phase A
Description: AQoL-8D provides a global utility score and comprised of 35 questions from which 8 dimensions (Independent Living, Life Satisfaction, Mental Health, Coping, Relationships, Self Worth, Pain, and Senses) are derived. Each of the 8 scales is calculated based on the answers to 3 questions. Each question is given an answer dependent utility score (0 [worst] to 1 [best]) and then these scores are combined using a multiplicative model to get the normalized scale score value, each scale ranging between 0.0 (representing death) and 1.0 (representing full health).
Time Frame: as for outcome 18
Population: FAS population. "Number Analyzed" = participants who were evaluable at the specified time point for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase A
Number analyzed (Participants) | 128
units on a scale
  Phase A Baseline: number analyzed (Participants) | 123
  Phase A Baseline | 0.747 (0.1819)
  Phase A Visit 2 (Weeks 8-9): number analyzed (Participants) | 100
  Phase A Visit 2 (Weeks 8-9) | 0.760 (0.1710)
  Phase A Visit 3 (Weeks 16-17): number analyzed (Participants) | 81
  Phase A Visit 3 (Weeks 16-17) | 0.767 (0.1691)
  Phase A Visit 4 (Weeks 24-25): number analyzed (Participants) | 61
  Phase A Visit 4 (Weeks 24-25) | 0.796 (0.1650)
  Phase A Visit 5 (Weeks 32-33): number analyzed (Participants) | 43
  Phase A Visit 5 (Weeks 32-33) | 0.800 (0.1762)
  Phase A Visit 6 (Weeks 40-41): number analyzed (Participants) | 28
  Phase A Visit 6 (Weeks 40-41) | 0.831 (0.1578)
  Phase A Visit 7 (Weeks 48-49): number analyzed (Participants) | 23
  Phase A Visit 7 (Weeks 48-49) | 0.818 (0.1455)
  Phase A Visit 8 (Weeks 56-57): number analyzed (Participants) | 18
  Phase A Visit 8 (Weeks 56-57) | 0.851 (0.1043)
  Phase A Visit 9 (Weeks 64-65): number analyzed (Participants) | 19
  Phase A Visit 9 (Weeks 64-65) | 0.822 (0.1304)
  Phase A Visit 10 (Weeks 72-73): number analyzed (Participants) | 15
  Phase A Visit 10 (Weeks 72-73) | 0.827 (0.1426)
  Phase A Visit 11 (Weeks 80-81): number analyzed (Participants) | 14
  Phase A Visit 11 (Weeks 80-81) | 0.839 (0.1272)
  Phase A Visit 12 (Weeks 88-89): number analyzed (Participants) | 14
  Phase A Visit 12 (Weeks 88-89) | 0.856 (0.1295)
  Phase A Visit 13 (Weeks 96-97): number analyzed (Participants) | 12
  Phase A Visit 13 (Weeks 96-97) | 0.831 (0.1482)
  Phase A Visit 14 (Weeks 104-105): number analyzed (Participants) | 12
  Phase A Visit 14 (Weeks 104-105) | 0.815 (0.1788)
  Phase A Visit 15 (Weeks 112-113): number analyzed (Participants) | 10
  Phase A Visit 15 (Weeks 112-113) | 0.871 (0.0877)
  Phase A Visit 16 (Weeks 120-121): number analyzed (Participants) | 8
  Phase A Visit 16 (Weeks 120-121) | 0.869 (0.1428)
  Phase A Visit 17 (Weeks 128-129): number analyzed (Participants) | 10
  Phase A Visit 17 (Weeks 128-129) | 0.859 (0.1430)
  Phase A Visit 18 (Weeks 136-137): number analyzed (Participants) | 9
  Phase A Visit 18 (Weeks 136-137) | 0.880 (0.1048)
  Phase A Visit 19 (Weeks 144-145): number analyzed (Participants) | 7
  Phase A Visit 19 (Weeks 144-145) | 0.915 (0.0883)
  Phase A Visit 20 (Weeks 152-153): number analyzed (Participants) | 7
  Phase A Visit 20 (Weeks 152-153) | 0.864 (0.1266)
  Phase A Visit 21 (Weeks 160-161): number analyzed (Participants) | 3
  Phase A Visit 21 (Weeks 160-161) | 0.806 (0.1422)
  Phase A Visit 22 (Weeks 168-169): number analyzed (Participants) | 2
  Phase A Visit 22 (Weeks 168-169) | 0.811 (0.2238)
  Phase A Visit 23 (Weeks 176-177): number analyzed (Participants) | 2
  Phase A Visit 23 (Weeks 176-177) | 0.709 (0.3336)
  Phase A EOT Visit (up to 4 years): number analyzed (Participants) | 80
  Phase A EOT Visit (up to 4 years) | 0.739 (0.1882)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 9
  Survival Follow-Up 1 (up to 4 years) | 0.718 (0.1600)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 2 (up to 4 years) | 0.792 (0.1977)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 2
  Survival Follow-Up 3 (up to 4 years) | 0.696 (0.1684)
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 0.620
  Survival Follow-Up 5 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 5 (up to 4 years) | 0.800
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 2
  Survival Follow-Up 6 (up to 4 years) | 0.810 (0.0531)
  Survival Follow-Up 7 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 7 (up to 4 years) | 0.874

20. Secondary Outcome: AQoL-8D Global Utility Score: Phase B
Description: AQoL-8D provides a global utility score and consists of 8 separately scored dimensions including Independent Living, Life Satisfaction, Mental Health, Coping, Relationships, Self Worth, Pain, and Senses. Each of the 8 scales is calculated based on the answers to 3 questions. Each question is given an answer dependent utility score (0 [worst] to 1 [best]) and then these scores are combined using a multiplicative model to get the normalized scale score value, each scale ranging between 0.0 (representing death) and 1.0 (representing full health).
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
units on a scale
  Phase B Baseline | 0.736 (0.1943)
  Phase B Visit 2 (up to 4 years): number analyzed (Participants) | 32
  Phase B Visit 2 (up to 4 years) | 0.773 (0.1821)
  Phase B Visit 3 (up to 4 years): number analyzed (Participants) | 23
  Phase B Visit 3 (up to 4 years) | 0.813 (0.1610)
  Phase B Visit 4 (up to 4 years): number analyzed (Participants) | 18
  Phase B Visit 4 (up to 4 years) | 0.878 (0.1154)
  Phase B Visit 5 (up to 4 years): number analyzed (Participants) | 13
  Phase B Visit 5 (up to 4 years) | 0.808 (0.1630)
  Phase B Visit 6 (up to 4 years): number analyzed (Participants) | 12
  Phase B Visit 6 (up to 4 years) | 0.809 (0.1717)
  Phase B Visit 7 (up to 4 years): number analyzed (Participants) | 6
  Phase B Visit 7 (up to 4 years) | 0.825 (0.1682)
  Phase B Visit 8 (up to 4 years): number analyzed (Participants) | 3
  Phase B Visit 8 (up to 4 years) | 0.910 (0.1023)
  Phase B Visit 9 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 9 (up to 4 years) | 0.819 (0.1986)
  Phase B Visit 10 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 10 (up to 4 years) | 0.856 (0.1589)
  Phase B Visit 11 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 11 (up to 4 years) | 0.730 (0.2906)
  Phase B Visit 12 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 12 (up to 4 years) | 0.960
  Phase B Visit 13 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 13 (up to 4 years) | 0.965
  Phase B Visit 14 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 14 (up to 4 years) | 0.958
  Phase B Visit 15 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 15 (up to 4 years) | 0.967
  Phase B Visit 16 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 16 (up to 4 years) | 0.942
  Phase B Visit 17 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 17 (up to 4 years) | 0.927
  Phase B Visit 18 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 18 (up to 4 years) | 0.931
  Phase B Visit 19 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 19 (up to 4 years) | 0.866
  Phase B Visit 20 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 20 (up to 4 years) | 0.887
  Phase B Visit 21 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 21 (up to 4 years) | 0.940
  Phase B Visit 22 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 22 (up to 4 years) | 0.919
  Phase B Visit 23 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 23 (up to 4 years) | 0.937
  Phase B Visit 24 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 24 (up to 4 years) | 0.950
  Phase B EOT Visit (up to 4 years): number analyzed (Participants) | 32
  Phase B EOT Visit (up to 4 years) | 0.708 (0.2229)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 1 (up to 4 years) | 0.788 (0.0895)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 4
  Survival Follow-Up 2 (up to 4 years) | 0.791 (0.1829)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 3 (up to 4 years) | 0.989
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 0.981
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 6 (up to 4 years) | 0.875

21. Secondary Outcome: Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Score: Phase A
Description: FACT-C is one part of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System, which comprehensively assesses the health-related QoL of cancer participants and participants with other chronic illnesses. It is composed of 27 items of the general version of the FACT-C as a general core QoL measure and has a disease-specific subscale containing 9 colorectal cancer-specific items. It consists of total 36 items, summarized to 5 subscales: physical well-being (7 items), functional well-being (7 items), social/family well-being (7 items); all 3 subscales range from 0 to 28, emotional well-being (6 items) range from 0 to 24, colorectal cancer subscale (9 items) range from 0 to 36; higher subscale score=better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. Total possible score range: 0 to 144. High scale score represents a better QoL.
Time Frame: as for outcome 18
Population: FAS population. "Number Analyzed" = participants who were evaluable at the specified time point for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase A
Number analyzed (Participants) | 128
units on a scale
  Phase A Baseline: number analyzed (Participants) | 121
  Phase A Baseline | 103.84 (16.615)
  Phase A Visit 2 (Weeks 8-9): number analyzed (Participants) | 98
  Phase A Visit 2 (Weeks 8-9) | 103.33 (16.065)
  Phase A Visit 3 (Weeks 16-17): number analyzed (Participants) | 78
  Phase A Visit 3 (Weeks 16-17) | 106.34 (15.318)
  Phase A Visit 4 (Weeks 24-25): number analyzed (Participants) | 61
  Phase A Visit 4 (Weeks 24-25) | 109.66 (15.038)
  Phase A Visit 5 (Weeks 32-33): number analyzed (Participants) | 43
  Phase A Visit 5 (Weeks 32-33) | 109.39 (16.727)
  Phase A Visit 6 (Weeks 40-41): number analyzed (Participants) | 30
  Phase A Visit 6 (Weeks 40-41) | 111.30 (16.420)
  Phase A Visit 7 (Weeks 48-49): number analyzed (Participants) | 23
  Phase A Visit 7 (Weeks 48-49) | 111.40 (13.506)
  Phase A Visit 8 (Weeks 56-57): number analyzed (Participants) | 17
  Phase A Visit 8 (Weeks 56-57) | 113.51 (10.777)
  Phase A Visit 9 (Weeks 64-65): number analyzed (Participants) | 19
  Phase A Visit 9 (Weeks 64-65) | 113.92 (12.239)
  Phase A Visit 10 (Weeks 72-73): number analyzed (Participants) | 15
  Phase A Visit 10 (Weeks 72-73) | 115.11 (15.473)
  Phase A Visit 11 (Weeks 80-81): number analyzed (Participants) | 14
  Phase A Visit 11 (Weeks 80-81) | 114.00 (13.230)
  Phase A Visit 12 (Weeks 88-89): number analyzed (Participants) | 14
  Phase A Visit 12 (Weeks 88-89) | 115.99 (12.844)
  Phase A Visit 13 (Weeks 96-97): number analyzed (Participants) | 12
  Phase A Visit 13 (Weeks 96-97) | 113.54 (12.298)
  Phase A Visit 14 (Weeks 104-105): number analyzed (Participants) | 12
  Phase A Visit 14 (Weeks 104-105) | 112.36 (15.443)
  Phase A Visit 15 (Weeks 112-113): number analyzed (Participants) | 10
  Phase A Visit 15 (Weeks 112-113) | 119.48 (11.542)
  Phase A Visit 16 (Weeks 120-121): number analyzed (Participants) | 7
  Phase A Visit 16 (Weeks 120-121) | 116.38 (15.214)
  Phase A Visit 17 (Weeks 128-129): number analyzed (Participants) | 9
  Phase A Visit 17 (Weeks 128-129) | 113.69 (17.816)
  Phase A Visit 18 (Weeks 136-137): number analyzed (Participants) | 9
  Phase A Visit 18 (Weeks 136-137) | 112.94 (16.931)
  Phase A Visit 19 (Weeks 144-145): number analyzed (Participants) | 7
  Phase A Visit 19 (Weeks 144-145) | 117.55 (10.397)
  Phase A Visit 20 (Weeks 152-153): number analyzed (Participants) | 7
  Phase A Visit 20 (Weeks 152-153) | 115.86 (13.120)
  Phase A Visit 21 (Weeks 160-161): number analyzed (Participants) | 3
  Phase A Visit 21 (Weeks 160-161) | 106.00 (20.664)
  Phase A Visit 22 (Weeks 168-169): number analyzed (Participants) | 2
  Phase A Visit 22 (Weeks 168-169) | 112.00 (26.870)
  Phase A Visit 23 (Weeks 176-177): number analyzed (Participants) | 2
  Phase A Visit 23 (Weeks 176-177) | 105.00 (36.770)
  Phase A EOT Visit (up to 4 years): number analyzed (Participants) | 79
  Phase A EOT Visit (up to 4 years) | 103.94 (17.429)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 9
  Survival Follow-Up 1 (up to 4 years) | 102.89 (18.086)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 2 (up to 4 years) | 104.00 (8.047)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 2
  Survival Follow-Up 3 (up to 4 years) | 105.50 (10.607)
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 109.00
  Survival Follow-Up 5 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 5 (up to 4 years) | 119.00
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 6 (up to 4 years) | 103.61 (4.945)
  Survival Follow-Up 7 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 7 (up to 4 years) | 115.00

22. Secondary Outcome: FACT-C Score: Phase B
Description: FACT-C is one part of the FACIT Measurement System, which comprehensively assesses the health-related QoL of cancer participants and participants with other chronic illnesses. It is composed of 27 items of the general version of the FACT-C as a general core QoL measure and has a disease-specific subscale containing 9 colorectal cancer-specific items. It consists of total 36 items, summarized to 5 subscales: physical well-being (7 items), functional well-being (7 items), social/family well-being (7 items); all 3 subscales range from 0 to 28, emotional well-being (6 items) range from 0 to 24, colorectal cancer subscale (9 items) range from 0 to 36; higher subscale score=better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. Total possible score range: 0 to 144. High scale score represents a better QoL.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab: Phase B
Number analyzed (Participants) | 53
units on a scale
  Phase B Baseline | 103.47 (18.284)
  Phase B Visit 2 (up to 4 years): number analyzed (Participants) | 30
  Phase B Visit 2 (up to 4 years) | 108.71 (17.387)
  Phase B Visit 3 (up to 4 years): number analyzed (Participants) | 25
  Phase B Visit 3 (up to 4 years) | 108.19 (16.541)
  Phase B Visit 4 (up to 4 years): number analyzed (Participants) | 19
  Phase B Visit 4 (up to 4 years) | 114.89 (14.467)
  Phase B Visit 5 (up to 4 years): number analyzed (Participants) | 13
  Phase B Visit 5 (up to 4 years) | 110.60 (15.592)
  Phase B Visit 6 (up to 4 years): number analyzed (Participants) | 12
  Phase B Visit 6 (up to 4 years) | 111.28 (14.121)
  Phase B Visit 7 (up to 4 years): number analyzed (Participants) | 6
  Phase B Visit 7 (up to 4 years) | 114.78 (12.640)
  Phase B Visit 8 (up to 4 years): number analyzed (Participants) | 3
  Phase B Visit 8 (up to 4 years) | 120.39 (9.007)
  Phase B Visit 9 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 9 (up to 4 years) | 108.08 (18.267)
  Phase B Visit 10 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 10 (up to 4 years) | 110.50 (17.678)
  Phase B Visit 11 (up to 4 years): number analyzed (Participants) | 2
  Phase B Visit 11 (up to 4 years) | 109.33 (19.328)
  Phase B Visit 12 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 12 (up to 4 years) | 125.00
  Phase B Visit 13 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 13 (up to 4 years) | 119.00
  Phase B Visit 14 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 14 (up to 4 years) | 117.00
  Phase B Visit 15 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 15 (up to 4 years) | 126.00
  Phase B Visit 16 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 16 (up to 4 years) | 123.00
  Phase B Visit 17 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 17 (up to 4 years) | 127.00
  Phase B Visit 18 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 18 (up to 4 years) | 126.00
  Phase B Visit 19 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 19 (up to 4 years) | 127.00
  Phase B Visit 20 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 20 (up to 4 years) | 126.00
  Phase B Visit 21 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 21 (up to 4 years) | 123.00
  Phase B Visit 22 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 22 (up to 4 years) | 124.00
  Phase B Visit 23 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 23 (up to 4 years) | 126.00
  Phase B Visit 24 (up to 4 years): number analyzed (Participants) | 1
  Phase B Visit 24 (up to 4 years) | 130.00
  Phase B EOT Visit (up to 4 years): number analyzed (Participants) | 33
  Phase B EOT Visit (up to 4 years) | 101.67 (19.023)
  Survival Follow-Up 1 (up to 4 years): number analyzed (Participants) | 3
  Survival Follow-Up 1 (up to 4 years) | 98.72 (20.024)
  Survival Follow-Up 2 (up to 4 years): number analyzed (Participants) | 4
  Survival Follow-Up 2 (up to 4 years) | 102.50 (17.705)
  Survival Follow-Up 3 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 3 (up to 4 years) | 126.33
  Survival Follow-Up 4 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 4 (up to 4 years) | 125.00
  Survival Follow-Up 6 (up to 4 years): number analyzed (Participants) | 1
  Survival Follow-Up 6 (up to 4 years) | 124.67

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to 4 years)
Description: FAS population.
Arm/Group | Bevacizumab: Phase A and Phase B
Serious Adverse Events (participants affected / at risk) | 86/128
Other Adverse Events (participants affected / at risk) | 128/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: Phase A and Phase B (N=128)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 3
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 6
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Neutropenic colitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Rectal perforation (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Catheter site pain (General disorders) | 1
Extravasation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 12
Cholecystitis acute (Hepatobiliary disorders) | 1
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Eyelid infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Muscle abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia streptococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Jugular vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: Phase A and Phase B (N=128)
Anaemia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Abdominal distension (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 40
Abdominal pain upper (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 51
Diarrhoea (Gastrointestinal disorders) | 70
Dyspepsia (Gastrointestinal disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 26
Mouth ulceration (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 87
Rectal haemorrhage (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 36
Toothache (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 80
Mucosal inflammation (General disorders) | 31
Non-cardiac chest pain (General disorders) | 8
Oedema peripheral (General disorders) | 14
Pyrexia (General disorders) | 12
Oral candidiasis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 20
Fall (Injury, poisoning and procedural complications) | 10
Weight decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 28
Dehydration (Metabolism and nutrition disorders) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Back pain (Musculoskeletal and connective tissue disorders) | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Dizziness (Nervous system disorders) | 13
Dysaesthesia (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 20
Headache (Nervous system disorders) | 24
Lethargy (Nervous system disorders) | 9
Neuropathy peripheral (Nervous system disorders) | 80
Paraesthesia (Nervous system disorders) | 26
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 25
Proteinuria (Renal and urinary disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 26
Dry skin (Skin and subcutaneous tissue disorders) | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 38
Rash (Skin and subcutaneous tissue disorders) | 21
Hypertension (Vascular disorders) | 23
Hypotension (Vascular disorders) | 7
Haemorrhoids (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.